CLINICAL TRIAL: NCT07063940
Title: Home-based EXercise and motivAtional Program Before and After Liver Transplantation: EXALT
Brief Title: Home-based EXercise and motivAtional Program Before and After Liver Transplantation
Acronym: EXALT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_20-065
Record Dates: First submitted 2025-06-11; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplant Surgery
Keywords: liver disease; quality of life; Liver transplant; Exercise and motivation
MeSH Terms: conditions — Liver Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Group 2 (Active Comparator): Patient exercise advice leaflet before and after LT.
  Interventions: Other: Patient exercise advice leaflet before and after LT.
- Group 1: Home-based exercise and motivation support programme (Experimental): Remotely-monitored home-based exercise and theory-based motivation support programme whilst on the LT waiting list (max. 12 months) through to 24 weeks post-LT.
  Interventions: Other: Home-based exercise and theory-based motivation support programme

INTERVENTIONS:
Other: Home-based exercise and theory-based motivation support programme — 1. A remotely-monitored personalised home-based exercise programme (HBEP) and
  2. An autonomous motivation enhancement programme, known as Empowering Physio, delivered to physiotherapists to support them in delivering the HBEP.
  Arms: Group 1: Home-based exercise and motivation support programme
Other: Patient exercise advice leaflet before and after LT. — Control
  Arms: Control: Group 2

SUMMARY:
Liver disease is the 3rd commonest cause of death in adults of working age and liver transplantation (LT) remains the only cure for liver failure. LT exerts a huge stress on the body and mind, especially in people who are already physically and mentally frail because of their liver disease. Investigators know that being physically frailty prior to surgery results in a longer hospital stay because of postoperative complications and contributes to 1 in 10 patients either dying whilst still on the waiting list or shortly after LT. Exercise is one of the most powerful medical therapies available, with numerous proven benefits to patients with diseases like diabetes, heart disease and cancer. Despite this, exercise is not currently used in patients with liver failure or recovering from LT, due to a lack of robust evidence. Exercise may have the potential to improve the lives of people with liver disease and reduce the side-effects of LT surgery. The current standard of care for NHS patients awaiting LT is an advice leaflet. Evidence-based exercise programmes around the time of transplantation do not exist. Only a few small studies have indicated that supervised, hospital-based exercise can improve physical function and quality of life. AIMS: Investigators aim to determine the effect of a home-based exercise and motivation-support programme in patients undergoing LT on their quality of life after surgery. Investigators would also like to understand if exercise results in improvements in intricate measures of physical fitness and muscle function that account for changes in quality of life, and how the motivation-support component of the intervention enhances uptake and ongoing engagement of exercise pre and post LT.

DETAILED DESCRIPTION:
Investigators intend to perform a clinical trial, in which patients will be randomly allocated to receive either the home-based exercise/motivation support programme (intervention group) or a patient advice leaflet (control group) whilst on the LT waiting list. The intervention will begin whilst patients are on the LT waiting list and end 6 months after LT. The intervention will consist of regular strength and endurance exercises, tailored to each patient's level of fitness. During clinic visits and via telephone calls a physiotherapist will provide motivational support throughout the exercise programme. The trial will involve recruiting 266 patients over two years from two LT hospitals in England. Investigators shall assess the effectiveness of the intervention by measuring quality of life before and after the study period in both groups of patients. The intervention will be deemed effective if quality of life scores are higher with the intervention than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or over)
* Patients listed for a cadaveric, primary LT at QEUHB or the RFH
* Being an out-patient at the time of baseline trial visit (consent)

Exclusion Criteria:

Patients listed for LT for any of the following reasons:

* super-urgent LT (according to the Kings College criteria)
* multi-organ transplantation (e.g. combined liver and kidney transplant)
* live-related donor LT
* re-graft LT

Patients with an inability to safely comply with the exercise intervention due to:

* severe hepatic encephalopathy (grade 3 or 4; or as judged by the clinical investigators)
* oxygen-dependent hepato-pulmonary syndrome

Patients without liver failure, including:

* liver cancer in the absence of cirrhosis
* polycystic liver disease
* rare metabolic/genetic conditions (e.g. glycogen storage disorders)

Refusal or lacks capacity to give informed consent to participate in the trial, at the point of study visit 1 (baseline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The physical component score (PCS) from the short form-36 version 2.0 (SF-36v2) health-related Quality of Life questionnaire | Baseline (visit 1, week 0) up to 24 weeks post-LT
  The primary outcome measure for this trial is the PCS from the SF-36v2 health-related QoL questionnaire at 24 weeks post LT. The SF-36v2 questionnaire includes 36 questions composed of eight multi-item scales, which reflect the impact of health problems on both the physical and mental condition of the patient.(A higher score reflects better quality of life. Two summary sub-scores can be calculated which are weighted combinations of the 8 scales, one to reflect the impact on physical function (PCS) and one to reflect the impact on psychological function, known as the mental component score (MCS).Scoring of the SF-36v2 questionnaire will based on the instructions provided in the SF-36v2 user's manual.

SECONDARY OUTCOMES:
Surgical complications -Comprehensive Complication Index (CCI): | LT up to 24 weeks post-LT
  The CCI is a well validated, reproducible tool in surgery and LT, which provides a 0-100 index (0=no complications, 100=death) using the frequency and grade (CTCAE grade) of surgical-related complications (i.e. wound dehiscence, bile leak, abdominal collections, bleeding, hepatic artery thrombosis etc).
Mental Component Score (MCS) of SF-36v2 health-related QoL questionnaire | Baseline (visit 1, week 0) up to 24 weeks post-LT
  The SF-36v2 questionnaire is a practical, reliable, and valid measure of physical and mental health that can be completed in 5 to 10 minutes. Scoring of the (MCS) SF-36v2 questionnaire is as described above for PCS SF-36v2 questionnaire.
Liver Frailty Index (LFI) | Baseline (visit 1, week 0) up to 24 weeks post-LT
  The LFI is a composite metric of three performance-based measures: hand grip strength (HGS), time to do 5 chair stands (seconds) and time holding 3 balance positions (feet side by side, semi-tandem and tandem) to objectively assess physical frailty in ambulatory patients with end-stage liver disease. The LFI score can be calculated using an on-line calculator (available at: http://liverfrailtyindex.ucsf.edu) with patient physical frailty categorised as robust, pre-frail and frail according to their index (index ≤ 3.2 (robust), 3.2-4.5 (pre-frail), >4.5 (frail)).
Duke activity status index (DASI): | Baseline (visit 1, week 0) up to 24 weeks post-LT
  The DASI is a 12 item self-reported assessment of functional capacity that requires minimal time to complete. It provides prognostic information in a variety of chronic diseases and can be used as an index of disease progression over time .
Pre-LT mortality (*assessed up to day of LT) | Baseline (visit 1, week 0) up to LT or the 48 week visit.
  The date and cause (based on death certificate) of death will be recorded.
Pre-LT UKELD | Baseline (visit 1, week 0) up to LT or the 48 week visit.
  UKELD: a scoring system (using a patient's international normalized ratio (INR), serum bilirubin, creatinine and sodium) used to predict the prognosis of patients with end-stage liver disease.
Pre-LT MELD-Na | Baseline (visit 1, week 0) up to LT or the 48 week visit.
  MELD-Na Score: is a scoring system created in 2008, based on the original MELD score, but with the addition of serum sodium. The MELD-Na, largely used for prioritisation in the United States, is a better predictor of mortality than the MELD score. Patients on oral anti-coagulants (including warfarin and the new oral anti-coagulants; predicted to be <2%) will be excluded from the analysis, as their UKELD/MELD-Na will be artificially high.
Pre-LT unscheduled hospitalisations | Baseline (visit 1, week 0) up to LT or the 48 week visit.
  Unscheduled hospital admissions: The frequency and duration (days) of non-elective hospital admissions .
Post-LT length of ICU stay (hours) | Between Liver transplant and immediately post-LT
  Length of ICU stay (hours)
length of hospital stay | Between Liver transplant and immediately post-LT
  length of hospital stay (days)
Re-listing for transplant | Between Liver transplant and Visit 9 (24 weeks post liver transplant)
  Re-listing for transplant will be recorded (date, reason) .
Post-LT mortality: | Between Liver transplant and Visit 10 (48 weeks post liver transplant)
  The date and cause (based on death certificate) of death will be recorded.
Habitual physical activity levels | Between Baseline (visit 1, week 0) and 24 weeks post LT
  Habitual (daily) levels of physical activity engagement (light, moderate and vigorous intensity) which may occur during the course of the trial will be measured using a 'blinded' wrist worn accelerometer (Actigraph GT9X). These will be worn for 14 days (24 hours/day):
  * Baseline (visit 1, week 0) to 14 days
  * 14 days before visit 2 (6 weeks), visit 3 (12 weeks) and visit 4 (24 weeks) pre-LT
  * 14 days before visit 7 (6 weeks post-LT), visit 8 (12 weeks post-LT) and visit 9 (24 weeks post-LT, end of intervention) Data captured during the 14-day periods will be analysed to quantify daily time (min/day) spent in; (1) light physical activity (1.6 - 2.9 metabolic equivalents (METS), (2) moderate physical activity (≥ 3 - 5.9 METS), (3) vigorous physical activity (≥6 METS), and sedentary time (≤1.5 METS).
"Dose" of exercise completed (measure of the frequency, intensity and duration of exercise) | Between Baseline ((visit 1, week 0) and 24 weeks post LT
  Data will be analysed from the 'blinded' wrist worn accelerometer (Actigraph GT9X) to understand the intensity and duration of the exercises completed during the 14 day periods.
Adherence to HBEP (intervention arm only) | Between study baseline (visit 1) and 24 weeks post LT
  Adherence to the HBEP will be measured using the 'blinded' wrist-worn accelerometer worn in the 14 day periods (described above). In addition, the participant will fill a self-reported exercise diary throughout the trial, which will be reviewed by the physiotherapist at each face-to-face trial visit until visit 9 (24 weeks post-LT, end of intervention). Using the diary, the physiotherapist will document how many structured HBEP sessions the participant has completed per week (maximum 5 per week).
Perceptions of the health care climate (how need supportive/empowering the physiotherapist is) | Between Baseline (visit 1, week 0) and 24 weeks post LT
  This will be measured using the Health Care Climate Questionnaire (HCCQ). The HCCQ comprises 15 items/statements which represent the patient's perceptions of the degree to which they feel their interactions with their physiotherapist (health care climate) empower them to engage in exercise (e.g. "I feel that my physiotherapist has provided me choices and options"). Patients are asked to respond to each item, indicating the extent to which they agree with each statement, on a Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Basic psychological need satisfaction (i.e. feelings of autonomy, relatedness, competence) | Between Baseline (visit 1, week 0) and 24 weeks post LT
  This will be measured using the Basic Psychological Need Satisfaction in Exercise Scale (PNSE): The PNSE will be used to examine participants basic psychological need satisfaction, in relation to their exercise engagement. The PNSE comprises 18 items, capturing the three basic psychological needs of autonomy (6 items, e.g. "I feel free to exercise in my own way"), competence (6 items, e.g. "feel that I am able to complete exercises that are personally challenging") and relatedness (6 items, e.g. I feel connected to the people who I interact with while I exercise"). Participants are asked to respond to each item, indicating the degree with which they agree with each statement, on a Likert scale from 1 (false) to 6 (true).
Self-determined motivation to exercise | Between Baseline (visit 1, week 0) and 24 weeks post LT
  This will be measured using the Behavioural Regulation in Exercise Questionaire-2 (BREQ-2). The BREQ-2 will measure participant's degree of self-determined motivation to engage in exercise, by assessing their external, introjected, identified and intrinsic regulations, as well as motivation. Following the stem, "I take part in exercise" participants will be asked to respond to 19 items assessing intrinsic regulation (4 items; e.g., "because I enjoy doing this"), identified regulation (4 items; e.g., "because I value the benefits of doing this"), introjected regulation (3 items; e.g., "because I feel guilty when I am not doing this"), external regulation (4 items; e.g., "because my friends and family say I should") and motivation (4 items; e.g., "but I think doing this is a waste of time"). Participants were asked to rate their agreement with each statement on a 5-point Likert scale from 0 (not true for me) to 4 (very true for me).

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Armstrong, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Birmingham Clinical Trials Unit (BCTU), Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — http://www.birmingham.ac.uk/ExaLT
- Available data/document: Study Protocol — http://www.birmingham.ac.uk/ExaLT
- Available data/document: Informed Consent Form — http://www.birmingham.ac.uk/ExaLT

DOCUMENTS (1):
  • Study Protocol (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT07063940/Prot_000.pdf